CLINICAL TRIAL: NCT04128228
Title: Neurobiological Responses in Alcoholism and Early Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000024809; 1R01AA026844 (NIH)
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Results first posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-10

CONDITIONS: Alcohol Use Disorder; Early Trauma Complications
Keywords: Alcohol use disorder; Early trauma; fMRI; Stress hormone; Alcohol relapse
MeSH Terms: conditions — Alcoholism; Wounds and Injuries | interventions — Ambulatory Care

STUDY DESIGN:
Intervention Model Description: Following baseline assessments including multimodal neuroimaging, AUD individuals with and without a history of early trauma received an equivalent 8-week outpatient treatment. Control participants with and without early trauma did not receive any treatment after baseline assessments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Alcohol use disorder with early trauma (Other): Individuals with alcohol use disorder participated in an equivalent 8-week outpatient treatment program.
  Interventions: Behavioral: 8-week outpatient treatment
- Alcohol use disorder without early trauma (Other): Individuals with alcohol use disorder participated in an equivalent 8-week outpatient treatment program.
  Interventions: Behavioral: 8-week outpatient treatment
- Controls with early trauma (No Intervention): Control participants did not receive any treatment.
- Controls without early trauma (No Intervention): Control participants did not receive any treatment.

INTERVENTIONS:
Behavioral: 8-week outpatient treatment — Individuals with AUD participated in an 8-week treatment program integrating cognitive behavioral techniques focused on emotion regulation with breathing-based stress management.
  Arms: Alcohol use disorder with early trauma; Alcohol use disorder without early trauma

SUMMARY:
Alcohol use disorder (AUD) accompanied by early trauma presents clinical challenges, including elevated rates of comorbid emotional symptoms and relapse. To better understand this co-occurring condition, this study investigates the neurobiological responses associated with AUD and early trauma. Using a multimodal neuroimaging approach, including functional magnetic resonance imaging (fMRI), the study concurrently measures brain activity and stress hormone responses in individuals with AUD and control participants, both with and without early trauma. The primary goal is to examine neurobiological responses and relapse patterns following treatment in individuals with AUD, with and without a history of early trauma. Conventional alcohol treatments often fail to specifically address the emotional complications in AUD individuals with early trauma. Therefore, this study also explores whether incorporating stress regulation into alcohol relapse prevention can improve outcomes for this population. Following baseline assessments that included multimodal neuroimaging, all participants with AUD received an 8-week outpatient treatment program integrating cognitive-behavioral methods focused on emotion regulation with stress reduction techniques, particularly self-regulated breathing strategies.

DETAILED DESCRIPTION:
The study recruited four demographically matched groups (age, sex ratio): individuals with AUD with and without a history of early trauma, and moderate drinkers with and without early trauma. Study procedures involved functional magnetic resonance imaging (fMRI), an eight-week outpatient treatment program, and a 90-day follow-up period. During fMRI sessions, participants engaged in a validated emotion provocation task, viewing stress, alcohol-cue, and neutral images while concurrent brain and stress hormone data are collected. Individuals with AUD completed baseline assessments, including multimodal neuroimaging, and then participated in an 8-week treatment program consisting of two sessions per week. This program integrated cognitive-behavioral techniques focused on emotion regulation with breathing-based stress management. Control participants completed baseline assessments including multimodal neuroimaging but did not receive any treatment. Following the treatment, participants with AUD were prospectively followed for 90 days, with remote follow-up interviews conducted at 14, 30, 90 days via video communication.

ELIGIBILITY:
AUD inclusion Criteria:

* Alcohol use disorder
* Either low or high early trauma (based on the Childhood Trauma Questionnaire)
* Body mass index (BMI) up to 35 (due to weight limitations of the MRI scanner)

AUD exclusion Criteria:

* Current or past substance use disorder other than alcohol; excluding caffeine and nicotine
* Psychiatric disorders except for mood and anxiety disorders
* Any significant current medical conditions
* Women who are peri- and post- menopausal, pregnant or lactating
* MRI specific exclusion criteria (e.g., claustrophobia, implanted metal in the body)

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dongju Seo, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited starting on October 3, 2019 through online platforms and flyers. A recruitment center was located in New Haven, Connecticut.
Pre-assignment Details: Out of the 148 enrolled participants, 17 individuals did not start the study due to participant withdrawal (N=14), MRI-day ineligibility (N=2), and non-compliance (N=1).
Groups:
- AUD/ET: Individuals with alcohol use disorder and early trauma:
  Individuals with alcohol use disorder will receive an 8-week outpatient treatment, involving two sessions per week that integrate cognitive behavioral therapy with breathing-based stress management.
- AUD/NT: Individuals with alcohol use disorder without early trauma:
  Individuals with alcohol use disorder will receive an 8-week outpatient treatment, involving two sessions per week that integrate cognitive behavioral therapy with breathing-based stress management.
- MD/ET: Moderate social drinkers (controls) with a history of early trauma: Control participants will undergo a baseline assessment without receiving any outpatient treatment.
- MD/NT: Moderate social drinkers (controls) without a history of early trauma: Control participants will undergo a baseline assessment without receiving any outpatient treatment.
Period: Overall Study
Arm/Group | AUD/ET | AUD/NT | MD/ET | MD/NT
Started | 34 | 33 | 27 | 37
Completed | 29 | 28 | 27 | 37
Not Completed | 5 | 5 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 0 | 0
Not completed — noncompliance | 2 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Out of the 148 enrolled participants, 17 participants did not start the study due to participant withdrawal (N=14), MRI-day ineligibility (N=2), and non-compliance (N=1).
Groups:
- AUD/ET: Individuals with alcohol use disorder (AUD) and early trauma (ET):
  Individuals with alcohol use disorder completed baseline assessments and then received an 8-week outpatient treatment that integrates alcohol treatment based on cognitive behavioral methods with breathing-based stress management.
- AUD/NT: Individuals with alcohol use disorder without early trauma:
  Individuals with alcohol use disorder completed baseline assessments and then received an 8-week outpatient treatment that integrates alcohol treatment based on cognitive behavioral methods with breathing-based stress management.
- MD/ET: Moderate drinkers (controls) with early trauma:
  Control participants completed baseline assessments without receiving any outpatient treatment.
- MD/NT: Moderate drinkers (controls) without early trauma:
  Control participants completed baseline assessments without receiving any outpatient treatment.
- Total: Total of all reporting groups
Arm/Group | AUD/ET | AUD/NT | MD/ET | MD/NT | Total
Number analyzed (Participants) | 34 | 33 | 27 | 37 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (9.0) | 35.94 (9.1) | 31.6 (7.5) | 32.0 (7.7) | 33.5 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 13 | 16 | 16 | 64
  Male | 15 | 20 | 11 | 21 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 7 | 12 | 32
  Not Hispanic or Latino | 28 | 26 | 20 | 25 | 99
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 0 | 2
  Asian | 3 | 1 | 5 | 3 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 6 | 6 | 8 | 30
  White | 17 | 24 | 10 | 21 | 72
  More than one race | 3 | 1 | 2 | 0 | 6
  Unknown or Not Reported | 1 | 1 | 2 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 34 | 33 | 27 | 37 | 131
Early Trauma Score [Mean (Standard Deviation); unit: units on a scale] — The Childhood Trauma Questionnaire (CTQ) is a 28-item self-report questionnaire designed to assess childhood trauma and maltreatment, consisting of five subscales: emotional abuse, physical abuse, sexual abuse, emotional neglect, and physical neglect. Each subscale is scored separately, and the sum of these scores provides a CTQ total score ranging from 25 to 125. Higher total scores indicate greater levels of self-reported childhood trauma exposure. The total CTQ scores are presented in this table.
  units on a scale | 60.2 (17.3) | 34.4 (6.2) | 63.3 (13.6) | 30.6 (5.8) | 46.0 (18.7)
Amount of alcohol consumption (weekly) [Mean (Standard Deviation); unit: alcohol drinks (weekly)] — The amount of weekly alcohol consumption was assessed using the Timeline Follow-Back (TLFB) method, a calendar-based self-report measure commonly used to track daily alcohol use. Participants recalled their drinking behavior using a calendar and reported both the days they consumed alcohol and the number of drinks consumed on each of those days.
  alcohol drinks (weekly) | 18.9 (15.8) | 19.6 (13.6) | 1.9 (2.1) | 2.2 (2.0) | 10.8 (13.6)
Days of alcohol consumption (weekly) [Mean (Standard Deviation); unit: days of alcohol use (weekly)] — The number of days of weekly alcohol consumption was assessed using the Timeline Follow-Back (TLFB) method, a calendar-based self-report measure commonly used to track daily alcohol use. Participants recalled their drinking behavior using a calendar and reported both the days they consumed alcohol and the number of drinks consumed on each of those days.
  days of alcohol use (weekly) | 4.0 (2.2) | 4.1 (2.0) | 0.9 (0.9) | 1.2 (1.0) | 2.6 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Brain Response
Description: Brain responses during the viewing of stress, alcohol-cue, and neutral images were examined using functional magnetic resonance imaging (fMRI) during an emotion provocation task. A regions of interest (ROI) analysis was conducted to assess brain activity in the right ventromedial prefrontal cortex (VmPFC, BA10), a region identified a priori. The VmPFC ROI was defined using the Yale-Brodmann atlas, and beta values were obtained using the BioImage Suite. The beta coefficient represents the extent to which a specific condition contributes to changes in the BOLD (Blood Oxygen Level Dependent) signal in a particular brain region. A positive beta in the vmPFC would indicate an increased vmPFC response, whereas a negative beta would indicate a decreased vmPFC response compared to baseline. The magnitude of the beta reflects the strength of this effect: a larger absolute value, (whether positive or negative), suggests a greater change in brain activation in response to the condition.
Time Frame: baseline
Population: In AUD/ET, one participant did not complete the fMRI part of the study, resulting in N=33 for brain response. Among them, one participant only completed alcohol cue condition due to discomfort with the MRI scan. In AUD/NT, two participants did not complete the fMRI part of the study, resulting in N=31. In MD/ET, one participant did not complete the stress condition. In MD/NET, one participant did not complete the alcohol condition, and two participants did not complete the stress condition.
Measure: Mean (Standard Deviation); unit: unitless
Groups:
- AUD/ET: Individuals with alcohol use disorder and early trauma:
  Individuals with alcohol use disorder completed baseline assessments, including multimodal neuroimaging, and then received an 8-week outpatient treatment that integrates alcohol treatment based on cognitive behavioral methods with breathing-based stress management.
- AUD/NT: Individuals with alcohol use disorder without early trauma:
  Individuals with alcohol use disorder completed baseline assessments, including multimodal neuroimaging, and then received an 8-week outpatient treatment that integrates alcohol treatment based on cognitive behavioral methods with breathing-based stress management.
- MD/ET: Moderate drinkers (controls) with early trauma:
  Control participants completed baseline assessments, including multimodal neuroimaging, without receiving any outpatient treatment.
- MD/NT: Moderate drinkers (controls) without early trauma:
  Control participants completed baseline assessments, including multimodal neuroimaging, without receiving any outpatient treatment.
Arm/Group | AUD/ET | AUD/NT | MD/ET | MD/NT
Number analyzed (Participants) | 33 | 31 | 27 | 37
unitless
  R. VmPFC response to stress cue: number analyzed (Participants) | 32 | 31 | 26 | 35
  R. VmPFC response to stress cue | .015 (.31) | .010 (.19) | -.013 (.19) | .08 (.19)
  R. VmPFC response to alcohol cue: number analyzed (Participants) | 33 | 31 | 27 | 36
  R. VmPFC response to alcohol cue | .071 (.33) | .058 (.19) | -.042 (.28) | .067 (.022)
  R. VmPFC response to neutral cue: number analyzed (Participants) | 32 | 31 | 27 | 37
  R. VmPFC response to neutral cue | .042 (.24) | .01 (.31) | -.091 (.30) | .017 (.22)
Statistical Analysis 1: Comparison: AUD/ET vs AUD/NT vs MD/ET vs MD/NT; A regions of interest (ROI) analysis was conducted to evaluate brain activity in the right ventromedial prefrontal cortex (VmPFC, BA10), a region identified a priori. The VmPFC ROI was defined using the Yale-Brodmann atlas in the BioImage Suite application, from which the beta value for the VmPFC ROI was obtained for a Linear Mixed Model analysis; Test type: Other — Single group: All individuals with alcohol use disorder received the same treatment. Brain responses were examined at baseline in individuals with alcohol use disorder (AUD) with and without early trauma (AUD/ET, AUD/NT), as well as in moderate drinkers (MD) with and without early trauma (MD/ET, MD/NT); p < 0.05, Linear Mixed Model — A 2 × 2 × 3 Linear Mixed Model was conducted with Early Trauma Group (ET, NT) and Drinking Group (AUD, MD) as between-subjects factors, and Condition (stress, alcohol, neutral) as the within-subjects factor; F value for the 2 X 2 Group Interaction = 5.5

2. Primary Outcome: Stress Hormone Response (Cortisol to ACTH Ratio)
Description: Cortisol to Adrenocorticotropic Hormone (ACTH) ratio indicates the relationship between cortisol secretion and ACTH stimulation at baseline.
  Cortisol is measured in micrograms per deciliter (µg/dL) and ACTH (adrenocorticotropic hormone) is measured in picograms per milliliter (pg/mL). Therefore, the unit of cortisol to ACTH ratio is expressed in µg/dL per pg/mL. Stress hormone samples were collected during the MRI scan.
Time Frame: baseline
Population: Among the 33 AUD/ET participants who underwent MRI scans, 3 blood samples were not collected due to nurse unavailability (N=2) and difficult venous access (N=1). In the 31 AUD/NT MRI participants, two samples were not collected due to technical issues. Of the 27 MD/ET, 5 samples were not collected due to nurse unavailability (N=5) and a technical issue (N=1). Of the 37 MD/NT, 6 samples were not collected due to nurse unavailability (N=4), IV tubing issue (N=1), and participant refusal (N=1).
Measure: Mean (Standard Deviation); unit: µg/dL per pg/ml
Groups:
- AUD/ET: Individuals with alcohol use disorder and early trauma:
  Individuals with alcohol use disorder completed baseline assessments including multimodal neuroimaging. Then, they participated in an 8-week outpatient treatment program integrating cognitive-behavioral techniques focused on emotion regulation with breathing-based stress management.
- AUD/NT: Individuals with alcohol use disorder without early trauma:
  Individuals with alcohol use disorder completed baseline assessments including multimodal neuroimaging. Then, they participated in an 8-week outpatient treatment program integrating cognitive-behavioral techniques focused on emotion regulation with breathing-based stress management.
- MD/ET: Moderate drinkers with early trauma:
  Control participants completed baseline assessments including multimodal neuroimaging but did not receive any treatment.
- MD/NT: Moderate drinkers without early trauma:
  Control participants completed baseline assessments including multimodal neuroimaging but did not receive any treatment.
Arm/Group | AUD/ET | AUD/NT | MD/ET | MD/NT
Number analyzed (Participants) | 29 | 29 | 22 | 31
µg/dL per pg/ml | .14 (.09) | .11 (.05) | .19 (.09) | .17 (.11)
Statistical Analysis 1: Comparison: AUD/ET vs AUD/NT vs MD/ET vs MD/NT; Test type: Other — Single group (all individuals with alcohol use disorder received the same treatment). Hormone responses were examined at baseline in individuals with alcohol use disorder (AUD) with and without early trauma (AUD/ET, AUD/NT), as well as in moderate drinkers (MD) with and without early trauma (MD/ET, MD/NT); p < 0.01, ANOVA; F value = 4.79

3. Primary Outcome: Time to Relapse
Description: The first day of alcohol consumption after treatment during the 90-day follow-up period. Alcohol use data was measured using the Timeline Follow-Back (TLFB) method, a calendar-based self-report tool to track alcohol use. Participants recalled their drinking behavior using a calendar and reported both the days they consumed alcohol and the number of drinks consumed on each of those days. Alcohol use data during the 90-day follow-up period is available only for the AUD/ET and AUD/NT groups, as the MD/ET and MD/NT groups had not initiated treatment.
Time Frame: up to 90 days
Population: Among the 34 AUD/ET participants, one dropped out before starting treatment, leaving 33 to begin the 8-week intervention. Of these, 29 completed the treatment and follow-up. Among the 33 AUD/NT participants, two dropped out before the treatment, leaving 31 who initiated the treatment. Of these, 28 completed the treatment and two lost to follow-up for this measure. The MD/ET and MD/NT groups did not start treatment therefore no data was collected for the MD groups.
Measure: Mean (Standard Deviation); unit: days to first drink after treatment
Groups:
- AUD/ET: Individuals with alcohol use disorder and early trauma:
  After completing an 8-week outpatient treatment, individuals with AUD were prospectively followed for 90 days. Remote follow-up interviews were conducted at 14, 30, and 90 days via video communication.
- AUD/NT: Individuals with alcohol use disorder without early trauma:
  After completing an 8-week outpatient treatment, individuals with AUD were prospectively followed for 90 days. Remote follow-up interviews were conducted at 14, 30, and 90 days via video communication.
Arm/Group | AUD/ET | AUD/NT
Number analyzed (Participants) | 29 | 26
days to first drink after treatment | 22.8 (34.0) | 5.6 (8.7)
Statistical Analysis 1: Comparison: AUD/ET vs AUD/NT; Test type: Other — Single Group; p < 0.05, Regression, Cox; Hazard Ratio (HR) = .71, 95% CI 2-sided [.53 to .95]

4. Secondary Outcome: Amount of Alcohol Consumption (Weekly)
Description: Average weekly alcohol consumption over the 90-day follow-up period. Alcohol use data was measured using the Timeline Follow-Back (TLFB) method, a calendar-based self-report tool to track alcohol use. Participants recalled their drinking behavior using a calendar and reported both the days they consumed alcohol and the number of drinks consumed on each of those days. Alcohol use data during the 90-day follow-up period is available only for the AUD/ET and AUD/NT groups, as the MD/ET and MD/NT groups had not initiated treatment.
Time Frame: up to 90 days
Population: Among the 34 AUD/ET participants, one dropped out before treatment, leaving 33 to start the intervention, with 29 completing treatment and follow-up (FU). Among the 33 AUD/NT participants, two dropped out before treatment, leaving 31 to initiate the intervention, with 28 completing treatment and three lost to follow-up for this measure (two before the 14-day FU, one before the 90-day FU). The MD/ET and MD/NT groups did not start treatment therefore no data was collected for the MD groups.
Measure: Mean (Standard Deviation); unit: alcohol drinks (weekly)
Arm/Group | AUD/ET | AUD/NT
Number analyzed (Participants) | 29 | 25
alcohol drinks (weekly) | 5.6 (8.1) | 13.1 (8.4)
Statistical Analysis 1: Comparison: AUD/ET vs AUD/NT; Test type: Other — Single Group. All individuals with alcohol use disorder received the same treatment; p < 0.01, t-test, 2 sided; t value = -3.35

5. Secondary Outcome: Frequency of Alcohol Use (Percentage)
Description: Percentage of alcohol use days over the 90-day follow-up period. Alcohol use data was measured using the Timeline Follow-Back (TLFB) method, a calendar-based self-report tool to track alcohol use. Participants recalled their drinking behavior using a calendar and reported both the days they consumed alcohol and the number of drinks consumed on each of those days. Alcohol use data during the 90-day follow-up period is available only for the AUD/ET and AUD/NT groups, as the MD/ET and MD/NT groups had not initiated treatment.
Time Frame: up to 90 days
Population: Among the 34 AUD/ET participants, one dropped out before treatment, leaving 33 to start the 8-week intervention, with 29 completing treatment and follow-up (FU). Among the 33 AUD/NT participants, two dropped out before treatment, leaving 31 to initiate the intervention, with 28 completing treatment and three lost to follow-up (two before the 14-day FU, one before the 90-day FU). The MD/ET and MD/NT groups did not start treatment therefore no data was collected for the MD groups.
Measure: Mean (Standard Deviation); unit: Percentage of alcohol use days
Groups:
- AUD/ET: Individuals with alcohol use disorder and early trauma:
  After receiving an 8-week outpatient treatment, AUD individuals were prospectively followed for 90 days. There were remote follow-up interviews at 14, 30, 90 days via video communication.
- AUD/NT: Individuals with alcohol use disorder without early trauma:
  After receiving an 8-week outpatient treatment, AUD individuals were prospectively followed for 90 days. There were remote follow-up interviews at 14, 30, 90 days via video communication.
Arm/Group | AUD/ET | AUD/NT
Number analyzed (Participants) | 29 | 25
Percentage of alcohol use days | 26.1 (29.4) | 45.4 (25.0)
Statistical Analysis 1: Comparison: AUD/ET vs AUD/NT; Test type: Other — Single Group (All individuals with alcohol use disorder received the same treatment.); p < 0.05, t-test, 2 sided; t value = -2.6

ADVERSE EVENTS:
Time Frame: 5.5 months for individuals with alcohol use disorder; 1.5 months for individuals without alcohol use disorder
Groups:
- MD/ET: Moderate drinkers (controls) with early trauma:
  Control participants completed baseline assessments including multimodal neuroimaging but did not receive any treatment.
- MD/NT: Moderate drinkers (controls) without early trauma:
  Control participants completed baseline assessments including multimodal neuroimaging but did not receive any treatment.
Arm/Group | AUD/ET | AUD/NT | MD/ET | MD/NT
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/33 | 0/27 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33 | 0/27 | 0/37
Other Adverse Events (participants affected / at risk) | 4/34 | 0/33 | 0/27 | 0/37
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AUD/ET (N=34) | AUD/NT (N=33) | MD/ET (N=27) | MD/NT (N=37)
low back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) — One participant reported a single episode of low back pain in week 4, while another participant reported two episodes in weeks 3 and 5. All episodes were attributed to a pre-existing condition and were unrelated to study participation.
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — One participant contracted COVID-19 in week 9 after treatment, while another participant was infected during week 5 of the treatment. Both cases were regarded as unrelated to study participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT04128228/Prot_SAP_ICF_001.pdf